CLINICAL TRIAL: NCT02240381
Title: Metabolic and CD4+ T Cell Dysregulation in Post-Transplant Diabetes Mellitus
Brief Title: Predicting Development of Diabetes Mellitus in Patients Undergoing Allogeneic Stem Cell Transplant
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding expired
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Brian Engelhardt, MD, Assistant Professor of Medicine, Hematologist/Oncologist, Principal Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: VICC BMT 1426; NCI-2014-01250 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA068485 (NIH)
Record Dates: First submitted 2014-08-28; First posted 2014-09-15 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Diabetes Mellitus; Malignant Neoplasm
MeSH Terms: conditions — Diabetes Mellitus; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (OGTT, euglycemic hyperinsulinemic clamp) (Experimental): Patients undergo OGTT and a standard 2-step euglycemic hyperinsulinemic clamp procedure prior to HCT. Patients then undergo repeat OGTT and a 2-step euglycemic hyperinsulinemic clamp procedure once after HCT between days 90-100.
  Interventions: Procedure: assessment of therapy complications; Other: laboratory biomarker analysis

INTERVENTIONS:
Procedure: assessment of therapy complications — During OGTT 75gm of glucose will be given followed by phlebotomy
Procedure: assessment of therapy complications — During clamp procedure tritiated glucose, D20, regular insulin will be given, followed by phlebotomy.
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This clinical trial studies the physiology and immunology of new-onset post-transplant diabetes mellitus in patients undergoing allogeneic stem cell transplantation. Oral glucose tolerance testing (OGTT), euglycemic hyperinsulinemic clamps, and immune assays will be used to define the mechanisms associated with abnormal glucose homeostasis following stem cell transplantation. Information from this clinical trial could be used to develop standardized screening procedures or to develop optimal treatment strategies for patients developing post-transplant diabetes mellitus.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether pre-transplant insulin resistance predicts for the development of new onset post-transplant diabetes mellitus (PTDM) in individuals without diabetes undergoing matched related donor (MRD) hematopoietic stem cell transplant (HCT).

II. To define the role of circulating tissue-specific Th1 cells in the development of PTDM.

III. To characterize the phenotype and function of circulating tissue-specific regulatory T cells (Tregs) in HCT recipients with or without PTDM.

OUTLINE:

Patients undergo OGTT and a standard 2-step euglycemic hyperinsulinemic clamp procedure prior to HCT. Patients then undergo repeat OGTT and a 2-step euglycemic hyperinsulinemic clamp procedure once after HCT between days 90-100.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing MRD allogeneic HCT
* DONOR: Donors undergoing stem cell collection for match related allogeneic stem cell transplant

Exclusion Criteria:

* Patients who have not received an allogeneic HCT
* Recent or current history of diabetes mellitus, defined as:1) diabetes therapy within 6 months of enrollment, or 2) fasting blood glucose at "pre-admit" (screening) visit >= 126 mg/dL
* Pregnancy or breastfeeding
* Unrelated donor, umbilical cord blood, mismatched, or haploidentical transplants
* Patients receiving T cell depletion or thymoglobulin as part of their transplant
* Patients on established, chronic corticosteroid therapy (> 5 mg /day of prednisone or prednisone equivalent) prior to transplant; established, chronic corticosteroid therapy is defined as daily dosing of > 5 mg/day of prednisone or prednisone equivalent for at least 2 weeks prior to the start of conditioning/chemotherapy or plans to continue pre-transplant corticosteroids (> 5 mg/day of prednisone or prednisone equivalent) indefinitely after transplantation
* Inability to give informed consent
* Any condition which, in the opinion of the investigator, might interfere with study objective
* Any reason which, in the opinion of the investigator, adds additional risk to the patient
* DONOR: Individuals not donating stem cells
* DONOR: Pregnancy or breastfeeding
* DONOR: Inability to give informed consent
* DONOR: Any condition which, in the opinion of the investigator, might interfere with study objective

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-11-20 (Actual); Primary Completion 2019-01-08 (Actual); Study Completion 2019-01-08 (Actual)

PRIMARY OUTCOMES:
Pre-transplant peripheral insulin sensitivity and glucose disposal as defined by the peripheral insulin sensitivity index among patients who do or do not go on to develop PTDM | Up to 21 days pre-transplant
  Patients will be followed for 100 days after transplant for development of diabetes. Wilcoxon rank sum test will be applied to compare the population mean difference between these two groups. Multivariable logistic regression will evaluate whether the peripheral insulin sensitivity index is an independent predictor of PTDM after adjusting for the following covariates: fasting C-peptide level, conditioning (ablative vs. reduced intensity), or acute graft-versus-host disease (GVHD) requiring steroids. The estimated odds ratio (OR) and 95% confidence interval of the OR will be provided to measure the effect of the association.
Ratio of circulating, gut-homing (alpha4beta7+) Th1 subsets pre-transplant with the development of PTDM after HCT | Up to day 100 after transplant
  Wilcoxon rank sum test will be applied to compare the mean difference between these two groups.
Expression of Helios or glycoprotein A repetitions predominant in alpha4beta7+Foxp3+ Tregs versus alpha4beta7+Foxp3- conventional T cells | Up to day 100 after transplant
  Wilcoxon rank sum test or two-sample t-test will be applied to compare the mean difference between two groups. Data will be presented using means and standard deviations for continuous variables, as well as percentage and frequency for categorical variables.

SECONDARY OUTCOMES:
Changes in hepatic insulin sensitivity among patients with or without established PTDM | Baseline to day 90 after transplant
  Comparison between two independent groups, e.g., with or without PTDM, will be carried out using either two-sample t-test or Wilcoxon rank sum test for continuous variables and Chi-square test or Fisher's exact test for categorical variables.
Changes in peripheral insulin sensitivity among patients with or without established PTDM | Baseline to day 90 after transplant
  Comparison between two independent groups, e.g., with or without PTDM, will be carried out using either two-sample t-test or Wilcoxon rank sum test for continuous variables and Chi-square test or Fisher's exact test for categorical variables.
Changes in OGTT results among patients with or without established PTDM | Baseline to day 90 after transplant
  Comparison between two independent groups, e.g., with or without PTDM, will be carried out using either two-sample t-test or Wilcoxon rank sum test for continuous variables and Chi-square test or Fisher's exact test for categorical variables.
Changes in hepatic insulin sensitivity in the entire cohort | Baseline to day 90 after transplant
  For the comparison of the changes between baseline and day+90 after transplant in the entire cohort, the mean difference will be compared with paired Student's t-test or Wilcoxon signed rank test for continuous variables and a McNemar's test for categorical variables.
Changes in peripheral insulin sensitivity in the entire cohort | Baseline to day 90 after transplant
  For the comparison of the changes between baseline and day+90 after transplant in the entire cohort, the mean difference will be compared with paired Student's t-test or Wilcoxon signed rank test for continuous variables and a McNemar's test for categorical variables.
Changes in OGTT results among patients in the entire cohort | Baseline to day 90 after transplant
  For the comparison of the changes between baseline and day+90 after transplant in the entire cohort, the mean difference will be compared with paired Student's t-test or Wilcoxon signed rank test for continuous variables and a McNemar's test for categorical variables.
Changes in hepatic insulin sensitivity among different groups | Baseline to day 90 after transplant
  To compare the differences between baseline (pre-transplant) and day +90 test results among various groups, linear mixed model will be applied to continuous outcomes (i.e., peripheral insulin sensitivity and hepatic glucose production) and generalized linear mixed model to noncontinuous outcomes (i.e., OGTT results). Groups of interest will be created by stratifying patients based on PTDM, conditioning regimen (ablative vs. reduced intensity) or acute GVHD treated with steroids.
Changes in peripheral insulin sensitivity among different groups | Baseline to day 90 after transplant
  To compare the differences between baseline (pre-transplant) and day +90 test results among various groups, linear mixed model will be applied to continuous outcomes (i.e., peripheral insulin sensitivity and hepatic glucose production) and generalized linear mixed model to noncontinuous outcomes (i.e., OGTT results). Groups of interest will be created by stratifying patients based on PTDM, conditioning regimen (ablative vs. reduced intensity) or acute GVHD treated with steroids.
Changes in OGTT results among different groups | Baseline to day 90 after transplant
  To compare the differences between baseline (pre-transplant) and day +90 test results among various groups, linear mixed model will be applied to continuous outcomes (i.e., peripheral insulin sensitivity and hepatic glucose production) and generalized linear mixed model to noncontinuous outcomes (i.e., OGTT results). Groups of interest will be created by stratifying patients based on PTDM, conditioning regimen (ablative vs. reduced intensity) or acute GVHD treated with steroids.
Ability of pre-transplant or post-transplant tissue-specific Tregs or Th1 cells to predict the development of PTDM | Up to day 100 after transplant
  The comparison between independent groups, e.g., with or without PTDM or the three OGTT groups (normal, impaired glucose tolerance, or diabetic), will be carried out using either Wilcoxon rank sum test or Kruskal-Wallis test, respectively.
Insulin clamp indices | Up to day 100 after transplant
  Spearman correlation will be used to evaluate the correlation between insulin clamp indices and Th1/Treg frequencies.
Th1/Treg frequencies | Up to day 100 after transplant
  Spearman correlation will be used to evaluate the correlation between insulin clamp indices and Th1/Treg frequencies.
Pre-HCT Th1 and Treg tissue-specific subsets | Up to 100 days pre-transplant
  Spearman correlation will evaluate the association between pre-HCT Th1 and Treg tissue-specific subsets with post-HCT donor derived Th1 and Treg.
Ability of alpha4beta7+ Tregs from patients with or without PTDM in suppressing the proliferation of allogeneic T cells | Up to day 90 after transplant
  Wilcoxon rank sum test or two-sample t-test will be applied to compare the mean difference between two groups. Data will be presented using means and standard deviations for continuous variables, as well as percentage and frequency for categorical variables. Investigations for outliers and assumptions for statistical analysis, e.g., normality and homoscedasticity will be made for the parametric test such as t-test and mixed model. If necessary, data will be transformed utilizing appropriate transformations such as the log or square root.
Ability of effector T cells from patients with PTDM to be resistant to suppression from Tregs obtained from healthy individuals | Up to day 100 after transplant
  Wilcoxon rank sum test or two-sample t-test will be applied to compare the mean difference between two groups. Data will be presented using means and standard deviations for continuous variables, as well as percentage and frequency for categorical variables.
Post-HCT donor derived Th1 and Treg subsets | Up to 100 days pre-transplant
  Spearman correlation will evaluate the association between pre-HCT Th1 and Treg tissue-specific subsets with post-HCT donor derived Th1 and Treg.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Engelhardt, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States